CLINICAL TRIAL: NCT03530826
Title: A Crowd Sourcing Platform for Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: All4Cure (Industry)
Responsible Party: Principal Investigator, Carl Anthony Blau, MD, Principal Investigator, All4Cure
Other Study IDs: All4Cure01
Record Dates: First submitted 2018-05-07; First posted 2018-05-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No Intervention

SUMMARY:
All4Cure aims to accelerate learning about cancer by sharing medical information and research results from cancer patients with fellow cancer patients, oncologists, and scientists on the All4Cure website with the hope that together patients, clinicians and researchers can cure cancer faster.

DETAILED DESCRIPTION:
The core hypothesis tested by this study is that engaging researchers, clinicians and patients in an online knowledge sharing platform will enable patients to better understand cancer, better inform treatment decisions made by oncologists and accelerate cancer research. Leftover samples from patients with cancer (blood, bodily fluids and/or tissues collected for clinical purposes) will be obtained and sent for various types of analyses and results will be shared on the All4Cure website.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with cancer.
* Be under the care of a physician.
* Be 18 years of age or older.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in tumor tissue molecular profiles | 6 years
  Profiles of pre- and post-treatment tumor tissue will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Blau, MD, Principal Investigator — All4Cure
Locations (1):
- All4Cure, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
nonidentifiable clinical and research data may be shared with other researchers.